CLINICAL TRIAL: NCT03051217
Title: Phase 2/3, Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study To Evaluate the Efficacy and Safety of Certolizumab Pegol in Japanese Subjects With Moderate to Severe Chronic Psoriasis
Brief Title: A Study to Test the Efficacy and Safety of Certolizumab Pegol in Japanese Subjects With Moderate to Severe Chronic Psoriasis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PS0017
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Results first posted 2019-12-11 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2020-11

CONDITIONS: Moderate to Severe Psoriasis; Generalized Pustular Psoriasis and Erythrodermic Psoriasis
Keywords: Psoriasis; PSO; Chronic plaque psoriasis; Certolizumb Pegol; Cimzia; Generalized pustular psoriasis and erythrodermic psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Certolizumab Pegol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo subcutaneous (sc) injection every two weeks (Q2W)
  Interventions: Other: Placebo
- CZP 200 mg (Experimental): Certolizumab Pegol subcutaneous (sc) injection 400 mg at Weeks 0, 2, 4, followed by Certolizumab Pegol subcutaneous (sc) injection 200 mg every two weeks (Q2W) with PBO administered to maintain the blind, starting at Week 6
  Interventions: Other: Placebo; Drug: Certolizumab Pegol
- CZP 400 mg (Experimental): Certolizumab Pegol subcutaneous (sc) injection 400 mg every two weeks (Q2W).
  Interventions: Drug: Certolizumab Pegol

INTERVENTIONS:
Other: Placebo — * Pharmaceutical Form: Solution for injection in pre-filled syringe
  * Concentration: 0.9 % saline
  * Route of Administration: Subcutaneous use Q2W
  Other Names: PBO
  Arms: CZP 200 mg; Placebo
Drug: Certolizumab Pegol — * Pharmaceutical Form: Solution for injection in pre-filled syringe
  * Concentration: 200 mg/mL
  * Route of Administration: Subcutaneous use
  Other Names: Cimzia; CDP870; CZP
  Arms: CZP 200 mg; CZP 400 mg

SUMMARY:
The purpose of this study is to demonstrate the efficacy and safety of Certolizumab Pegol (CZP) in the treatment of moderate to severe chronic plaque Psoriasis (PSO) in Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female, >= 20 years of age.
* Institutional Review Board-approved written informed consent form is signed and dated by the subject.
* Other protocol-defined inclusion criteria may apply.

For subjects with moderate to severe chronic plaque psoriasis (PSO)

* Chronic plaque psoriasis for at least 6 months.
* Baseline Psoriasis Activity and Severity Index (PASI) >=12 and Body Surface Area (BSA) affected by PSO >=10% and Physician's Global Assessment (PGA) score of 3 or higher.
* Candidates for systemic PSO therapy and/or phototherapy and/or chemophototherapy.

For subjects with generalized pustular PSO or erythrodermic PSO

* Diagnosis of generalized pustular PSO or erythrodermic PSO at Screening.
* History of plaque-type PSO if subjects have a diagnosis of erythrodermic PSO.
* Baseline BSA affected by PSO >=80% if subjects have a diagnosis of erythrodermic PSO.

Exclusion Criteria:

* Female subject who is breastfeeding, pregnant, or plans to become pregnant during the study or within 5 months following last dose of study drug. Male subject who is planning a partner pregnancy during the study or within 5 months following the last dose of study drug.
* Subject has guttate psoriasis or drug-induced psoriasis. For subjects with moderate to severe plaque psoriasis, erythrodermic or pustular forms of psoriasis also are excluded.
* History of current, chronic, or recurrent infections of viral, bacterial, or fungal origin as described in the protocol. Also, subjects with a high risk of infection in the Investigator's opinion.
* History of a lymphoproliferative disorder including lymphoma or current signs and symptoms suggestive of lymphoproliferative disease.
* History of other malignancy or concurrent malignancy as described in the protocol.
* Class III or IV congestive heart failure
* History of, or suspected, demyelinating disease of the central nervous system (e.g., multiple sclerosis or optic neuritis).
* Subject has any other condition which, in the Investigator's judgment, would make the subject unsuitable for inclusion in the study.
* Concurrent medication restrictions as described in the protocol.
* Subject with known tuberculosis (TB) infection, at high risk of acquiring TB infection, or with untreated latent tuberculosis infection (LTBI) or current or history of nontuberculous mycobacterial (NTMB) infection.
* Subject has any protocol defined clinically significant laboratory abnormalities at the screening
* Other protocol-defined exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2019-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — UCB (+1 844 599 2273)
Locations (33):
- Japan (33):
  - Ps0017 024, Asahikawa
  - Ps0017 012, Bunkyō City
  - Ps0017 010, Chiyoda-Ku
  - Ps0017 007, Chūōku
  - Ps0017 004, Fukuoka
  - Ps0017 039, Fukushima
  - Ps0017 028, Gifu
  - Ps0017 040, Hamamatsu
  - Ps0017 013, Itabashi-Ku
  - Ps0017 022, Kobe
  - Ps0017 032, Kumamoto
  - Ps0017 031, Kurume
  - Ps0017 021, Kyoto
  - Ps0017 041, Matsumoto
  - Ps0017 009, Minatoku
  - Ps0017 033, Miyazaki
  - Ps0017 016, Nagoya
  - Ps0017 029, Nankoku
  - Ps0017 005, Obihiro
  - Ps0017 017, Osaka
  - Ps0017 042, Osaka
  - Ps0017 037, Ōsaka-sayama
  - Ps0017 001, Sapporo
  - Ps0017 027, Sendai
  - Ps0017 015, Shimotsuke
  - Ps0017 008, Shinagawa-Ku
  - Ps0017 002, Shinjuku
  - Ps0017 003, Shinjuku
  - Ps0017 011, Shinjuku
  - Ps0017 014, Shinjuku
  - Ps0017 034, Sumida City
  - Ps0017 038, Takaoka
  - Ps0017 025, Tsu

REFERENCES:
- [Result] Imafuku S, Tada Y, Umezawa Y, Sakurai S, Hoshii N, Nakagawa H. Certolizumab Pegol in Japanese Patients with Moderate to Severe Plaque Psoriasis: Effect of Demographics and Baseline Disease Characteristics on Efficacy. Dermatol Ther (Heidelb). 2022 Jan;12(1):121-135. doi: 10.1007/s13555-021-00645-2. Epub 2021 Nov 26. PMID 34826124
- [Derived] Okubo Y, Umezawa Y, Sakurai S, Hoshii N, Nakagawa H. Efficacy and Safety of Certolizumab Pegol in Japanese Patients with Generalized Pustular Psoriasis and Erythrodermic Psoriasis: 52-Week Results. Dermatol Ther (Heidelb). 2022 Jun;12(6):1397-1415. doi: 10.1007/s13555-022-00741-x. Epub 2022 May 27. PMID 35622315
- [Derived] Umezawa Y, Asahina A, Imafuku S, Tada Y, Sano S, Morita A, Sakurai S, Hoshii N, Tilt N, Nakagawa H. Efficacy and Safety of Certolizumab Pegol in Japanese Patients with Moderate to Severe Plaque Psoriasis: 52-Week Results. Dermatol Ther (Heidelb). 2021 Jun;11(3):943-960. doi: 10.1007/s13555-021-00520-0. Epub 2021 Apr 22. PMID 33886085
- [Derived] Umezawa Y, Sakurai S, Hoshii N, Nakagawa H; PS0017 Study Group. Certolizumab Pegol for the Treatment of Moderate to Severe Plaque Psoriasis: 16-Week Results from a Phase 2/3 Japanese Study. Dermatol Ther (Heidelb). 2021 Apr;11(2):513-528. doi: 10.1007/s13555-021-00494-z. Epub 2021 Feb 19. PMID 33606269
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in February 2017 and concluded in January 2019.
Pre-assignment Details: The study included a 5 Week Screening Period, an Initial Period up to Week 16, a Maintenance Period up to Week 52 and a Safety Follow-up Period up to Week 60.
  Participant Flow refers to the Randomized Set (RS)
Groups:
- Placebo: This arm consisted of participants who received Placebo subcutaneous (sc) injection every two weeks (Q2W) during the Initial Period.
- CZP 200 mg Q2W: This arm consisted of participants who received Certolizumab Pegol (CZP) subcutaneous (sc) injection 400 mg at Weeks 0, 2, 4, followed by Certolizumab Pegol subcutaneous (sc) injection 200 mg every two weeks (Q2W) starting at Week 6 during the Initial Period.
- CZP 400 mg Q2W: This arm consisted of participants who received Certolizumab Pegol (CZP) subcutaneous (sc) injection 400 mg every two weeks (Q2W) during the Initial Period.
- Placebo/Placebo: This arm consisted of participants who were initially randomized to Placebo during the Initial Period, who achieved a PASI50 response at Week 16 and continued to receive Placebo during the Maintenance Period. Participants who did not achieve a PASI50 response at Week 16 escaped from the double-blind treatment and received open-label CZP 400 mg Q2W as 3 loading doses followed by CZP 200 mg Q2W.
- CZP 400 mg Q2W/CZP 400 mg Q2W: This arm consisted of participants who were initially randomized to CZP 400 mg Q2W during the Initial Period, who achieved a PASI50 response at Week 16 and continued to receive CZP 400 mg Q2W during the Maintenance Period. Participants who did not achieve a PASI50 response at Week 16 escaped from the double-blind treatment and received open-label CZP 400 mg Q2W as 3 loading doses followed by CZP 200 mg Q2W.
- CZP 200 mg Q2W/CZP 200 mg Q2W: This arm consisted of participants who were initially randomized to CZP 200 mg Q2W during the Initial Period, who achieved a PASI50 response at Week 16 and were re-randomized to receive CZP 200 mg Q2W during the Maintenance Period. Participants who did not achieve a PASI50 response at Week 16 escaped from the double-blind treatment and received open-label CZP 400 mg Q2W as 3 loading doses followed by CZP 200 mg Q2W.
- CZP 200 mg Q2W/CZP 400 mg Q4W: This arm consisted of participants who were initially randomized to CZP 200 mg Q2W during the Initial Period, who achieved a PASI50 response at Week 16 and were re-randomized to receive CZP 400 mg Q4W, with Placebo administered on alternate dosing weeks to maintain the blind, during the Maintenance Period. Participants who did not achieve a PASI50 response at Week 16 escaped from the double-blind treatment and received open-label CZP 400 mg Q2W as 3 loading doses followed by CZP 200 mg Q2W.
Period: Initial Period (Week 0 to Week 16)
Arm/Group | Placebo | CZP 200 mg Q2W | CZP 400 mg Q2W | Placebo/Placebo | CZP 400 mg Q2W/CZP 400 mg Q2W | CZP 200 mg Q2W/CZP 200 mg Q2W | CZP 200 mg Q2W/CZP 400 mg Q4W
Started | 26 | 48 | 53 | 0 | 0 | 0 | 0
Completed | 23 | 46 | 51 | 0 | 0 | 0 | 0
Not Completed | 3 | 2 | 2 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0 | 0 | 0 | 0
Period: Maintenance Period (Week 16 to Week 52)
Arm/Group | Placebo | CZP 200 mg Q2W | CZP 400 mg Q2W | Placebo/Placebo | CZP 400 mg Q2W/CZP 400 mg Q2W | CZP 200 mg Q2W/CZP 200 mg Q2W | CZP 200 mg Q2W/CZP 400 mg Q4W
Started | 0 | 0 | 0 | 23 | 51 | 26 | 20
Received Escape Treatment | 0 | 0 | 0 | 21 | 3 | 7 | 3
Completed | 0 | 0 | 0 | 20 | 48 | 24 | 19
Not Completed | 0 | 0 | 0 | 3 | 3 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 2 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Difficulty in going to hospital | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set which consisted of all participants in the Randomized Set (RS) who received at least 1 dose of study medication.
Arm/Group | Placebo | CZP 200 mg Q2W | CZP 400 mg Q2W | Total Title
Number analyzed (Participants) | 26 | 48 | 53 | 127
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 40 | 49 | 113
  >=65 years | 2 | 8 | 4 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.93 (11.37) | 48.43 (13.47) | 52.43 (11.59) | 50.00 (12.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 12 | 11 | 28
  Male | 21 | 36 | 42 | 99
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian (Japanese only) | 26 | 48 | 53 | 127

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving a 75 % or Higher Improvement in Psoriasis Area and Severity Index (PASI) Score at Week 16
Description: The PASI75 response assessments were based on at least 75 % improvement in the PASI score from Baseline. This is a scoring system that averages the redness, thickness, and scaliness of the psoriatic lesions (on a 0-4 scale), and weights the resulting score by the area of skin involved. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Time Frame: Week 16
Population: The Full Analysis Set (FAS) consisted of all participants in the Randomized Set (RS) who received at least 1 dose of the study medication and had valid efficacy assessments for Baseline and for at least 1 post-Baseline visit.
  Missing data were handled using the Markov Chain Monte Carlo (MCMC) method for multiple imputation.
Measure: Number; unit: percentage of participants
Groups:
- Placebo (FAS): This arm consisted of participants who received Placebo subcutaneous (sc) injection every two weeks (Q2W) during the Initial Period. Participants formed the Full Analysis Set (FAS).
- CZP 200 mg Q2W (FAS): This arm consisted of participants who received Certolizumab Pegol (CZP) subcutaneous (sc) injection 400 mg at Weeks 0, 2, 4, followed by Certolizumab Pegol subcutaneous (sc) injection 200 mg every two weeks (Q2W) starting at Week 6 during the Initial Period. Participants formed the FAS.
- CZP 400 mg Q2W (FAS): This arm consisted of participants who received Certolizumab Pegol (CZP) subcutaneous (sc) injection 400 mg every two weeks (Q2W) during the Initial Period. Participants formed the FAS.
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS) | CZP 400 mg Q2W (FAS)
Number analyzed (Participants) | 26 | 48 | 53
percentage of participants | 7.9 | 73.0 | 87.1
Statistical Analysis 1: Comparison: Placebo (FAS) vs CZP 200 mg Q2W (FAS); The primary and secondary efficacy endpoints were evaluated using a fixed-sequence testing procedure to account for multiplicity; Test type: Superiority; Regression, Logistic; If there is a group without a responder, in this case the biological exposure will be excluded from the model, an exact logistic regression applied; Estimated difference in responder rate = 65.1, 95% CI 2-sided [48.22 to 81.90] — If there is a group without a responder, in this case the biological exposure will be excluded from the model, an exact logistic regression applied
Statistical Analysis 2: Comparison: Placebo (FAS) vs CZP 400 mg Q2W (FAS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Estimated difference in responder rate = 79.1, 95% CI 2-sided [65.10 to 93.17] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo (FAS) vs CZP 200 mg Q2W (FAS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic — The p-value for the primary analysis was evaluated at a 2-sided significance level of 0.025 for each CZP dose vs PBO; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 31.695, 97.5% CI 2-sided [5.129 to 195.877]
Statistical Analysis 4: Comparison: Placebo (FAS) vs CZP 400 mg Q2W (FAS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic — The p-value for the primary analysis was evaluated at a 2-sided significance level of 0.025 for each CZP dose vs PBO; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 79.112, 97.5% CI 2-sided [11.739 to 533.168]

2. Secondary Outcome: Percentage of Subjects Who Achieve a Physician's Global Assessment (PGA) Clear or Almost Clear Response (With at Least 2-category Improvement) at Week 16
Description: This Outcome Measure applied to participants with moderate to severe chronic plaque Psoriasis (PSO).
  The Investigator assessed the overall severity of Psoriasis (PSO) using the following 5-point scale: 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe.
Time Frame: Week 16
Population: The Full Analysis Set (FAS) consisted of all participants in the RS who received at least 1 dose of the study medication and had valid efficacy assessments for Baseline and for at least 1 post-Baseline visit.
  Missing data were handled using the Markov Chain Monte Carlo (MCMC) method for multiple imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS) | CZP 400 mg Q2W (FAS)
Number analyzed (Participants) | 26 | 48 | 53
percentage of participants | 0.0 | 52.7 | 66.7
Statistical Analysis 1: Comparison: Placebo (FAS) vs CZP 200 mg Q2W (FAS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Estimated difference in responder rate = 52.7, 95% CI 2-sided [29.95 to 75.39] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo (FAS) vs CZP 400 mg Q2W (FAS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Estimated difference in responder rate = 66.7, 95% CI 2-sided [43.34 to 90.15] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo (FAS) vs CZP 200 mg Q2W (FAS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic — The p-value for the primary analysis was evaluated at a 2-sided significance level of 0.025 for each CZP dose vs PBO; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 38.193, 97.5% CI 2-sided [6.113 to 238.619]
Statistical Analysis 4: Comparison: Placebo (FAS) vs CZP 400 mg Q2W (FAS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic — The p-value for the primary analysis was evaluated at a 2-sided significance level of 0.025 for each CZP dose vs PBO; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 69.580, 97.5% CI 2-sided [11.138 to 434.659]

3. Secondary Outcome: Percentage of Subjects Achieving a 90 % or Higher Improvement in Psoriasis Area and Severity Index (PASI) Score at Week 16
Description: The PASI90 response assessments were based on at least 90 % improvement in the PASI score from Baseline. This is a scoring system that averages the redness, thickness, and scaliness of the psoriatic lesions (on a 0-4 scale), and weights the resulting score by the area of skin involved. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS) | CZP 400 mg Q2W (FAS)
Number analyzed (Participants) | 26 | 48 | 53
percentage of participants | 0.2 | 53.8 | 75.7
Statistical Analysis 1: Comparison: Placebo (FAS) vs CZP 200 mg Q2W (FAS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Estimated difference in responder rate = 53.6, 95% CI 2-sided [30.67 to 76.47] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo (FAS) vs CZP 400 mg Q2W (FAS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Estimated difference in responder rate = 75.5, 95% CI 2-sided [51.95 to 99.04] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo (FAS) vs CZP 200 mg Q2W (FAS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic — The p-value for the primary analysis was evaluated at a 2-sided significance level of 0.025 for each CZP dose vs PBO; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 38.696, 97.5% CI 2-sided [6.047 to 247.634]
Statistical Analysis 4: Comparison: Placebo (FAS) vs CZP 400 mg Q2W (FAS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic — The p-value for the primary analysis was evaluated at a 2-sided significance level of 0.025 for each CZP dose vs PBO; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 100.459, 97.5% CI 2-sided [15.540 to 649.437]

4. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) at Week 16
Description: This Outcome Measure applied to participants with moderate to severe chronic plaque Psoriasis (PSO).
  The DLQI is a subject-reported questionnaire designed for use in adult participants with PSO.
  The DLQI is a skin disease-specific questionnaire aimed at the evaluation of how symptoms and treatment affect patients' health related quality of life (HRQoL). This instrument asked participants about symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. It has been shown to be valid and reproducible in PSO patients. The DLQI score ranges from 0 to 30 with higher scores indicating lower HRQoL. A higher than or equal to (>=) 4-point change in the DLQI score (DLQI response) has been reported to be meaningful for the patient (within-patient minimal important difference Basra et al, 2015) a DLQI absolute score of lower than or equal to (=<) 1 indicates DLQI remission (i.e., no or small impact of the disease on HRQoL).
Time Frame: Baseline and Week 16
Population: The Full Analysis Set (FAS) consisted of all participants in the RS who received at least 1 dose of the study medication and had valid efficacy assessments for Baseline and for at least 1 post-Baseline visit.
  Missing data were handled using the last observation carried forward (LOCF) method for the DLQI.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS) | CZP 400 mg Q2W (FAS)
Number analyzed (Participants) | 26 | 48 | 53
Scores on a scale | -0.3 (1.0) | -6.8 (0.7) | -6.8 (0.7)
Statistical Analysis 1: Comparison: Placebo (FAS) vs CZP 200 mg Q2W (FAS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — p-value obtained for each treatment group comparison tested at a significance level of 0.025 in the fixed sequence testing procedure; ANCOVA model of change from Baseline DLQI score with treatment group and prior biologic exposure as factors and Baseline DLQI score as a covariate; Adjusted Mean Treatment Difference = -6.5, 97.5% CI 2-sided [-9.100 to -3.844]
Statistical Analysis 2: Comparison: Placebo (FAS) vs CZP 400 mg Q2W (FAS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 4, analysis 1]; Adjusted Mean Treatment Difference = -6.5, 97.5% CI 2-sided [-9.099 to -3.910]

5. Secondary Outcome: Change From Baseline in Itch Numeric Rating Scale at Week 16
Description: This Outcome Measure applied to participants with moderate to severe chronic plaque Psoriasis (PSO).
  The Itch Numeric Rating Scale (NRS) has been developed as a simple, single item instrument to assess the patient-reported severity of itch at its most intense during the past 24h period. Participants indicate itch severity by circling the integer that best describes the worst level of itching due to PSO in the past 24h period on an 11-point scale anchored at 0, representing "no itching" and 10, representing "worst itch imaginable" (Kimball et al, 2016).
Time Frame: Baseline and Week 16
Population: The Full Analysis Set (FAS) consisted of all participants in the RS who received at least 1 dose of the study medication and had valid efficacy assessments for Baseline and for at least 1 post-Baseline visit.
  Missing data were handled using the last observation carried forward (LOCF) method for the Itch Numeric Rating Scale.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS) | CZP 400 mg Q2W (FAS)
Number analyzed (Participants) | 26 | 48 | 53
Scores on a scale | 0.2 (0.5) | -2.9 (0.4) | -4.0 (0.3)
Statistical Analysis 1: Comparison: Placebo (FAS) vs CZP 200 mg Q2W (FAS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 4, analysis 1]; ANCOVA model of change from Baseline Itch NRS with treatment group and prior biologic exposure as factors and Baseline Itch NRS as a covariate; Adjusted Mean Treatment Difference = -3.1, 95% CI 2-sided [-4.265 to -2.002]
Statistical Analysis 2: Comparison: Placebo (FAS) vs CZP 400 mg Q2W (FAS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 5, analysis 1]; Adjusted Mean Treatment Difference = -4.2, 95% CI 2-sided [-5.295 to -3.069]

6. Secondary Outcome: Plasma Concentration of Certolizumab Pegol (CZP)
Description: Plasma concentration was expressed in micrograms per milliliter (μg/mL).
  Values below Lower Limit of Quantification (LLOQ) were set to half the LLOQ to present summaries.
  The geometric mean and geometric coefficient of variation were only displayed if at least 2/3 of the data were above the LLOQ.
Time Frame: Blood samples were collected at Baseline (Week 0) and at Weeks 2, 4, 6, 8, 12, 16, 24, 32, 40, 52, 60
Population: The Pharmacokinetics Per-Protocol Set (PK-PPS) consisted of all participants in the RS who took at least 1 dose of the study medication and provided at least 1 quantifiable CZP plasma concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- CZP 200 mg Q2W/CZP 200 mg Q2W (PK-PPS): This arm consisted of participants who were initially randomized to CZP 200 mg Q2W during the Initial Period, who achieved a PASI50 response at Week 16 and were re-randomized to receive CZP 200 mg Q2W during the Maintenance Period. Participants who did not achieve a PASI50 response at Week 16 escaped from the double-blind treatment and received open-label CZP 400 mg Q2W as 3 loading doses followed by CZP 200 mg Q2W. Participants formed the Pharmacokinetics Per-Protocol Set (PK-PPS).
- CZP 400 mg Q2W/CZP 400 mg Q2W (PK-PPS): This arm consisted of participants who were initially randomized to CZP 400 mg Q2W during the Initial Period, who achieved a PASI50 response at Week 16 and continued to receive CZP 400 mg Q2W during the Maintenance Period. Participants who did not achieve a PASI50 response at Week 16 escaped from the double-blind treatment and received open-label CZP 400 mg Q2W as 3 loading doses followed by CZP 200 mg Q2W. Participants formed the PK-PPS.
- CZP 200 mg Q2W/CZP 400 mg Q4W (PK-PPS): This arm consisted of participants who were initially randomized to CZP 200 mg Q2W during the Initial Period, who achieved a PASI50 response at Week 16 and were re-randomized to receive CZP 400 mg Q4W, with Placebo administered on alternate dosing weeks to maintain the blind, during the Maintenance Period. Participants who did not achieve a PASI50 response at Week 16 escaped from the double-blind treatment and received open-label CZP 400 mg Q2W as 3 loading doses followed by CZP 200 mg Q2W. Participants formed the PK-PPS.
Arm/Group | CZP 200 mg Q2W/CZP 200 mg Q2W (PK-PPS) | CZP 400 mg Q2W/CZP 400 mg Q2W (PK-PPS) | CZP 200 mg Q2W/CZP 400 mg Q4W (PK-PPS)
Number analyzed (Participants) | 28 | 53 | 20
µg/mL
  Baseline | NA (NA) — Values were below the level of detection. | NA (NA) — Values were below the level of detection. | NA (NA) — Values were below the level of detection.
  Week 2 | 34.6417 (28.3) | 35.2588 (25.2) | 33.2026 (26.0)
  Week 4: number analyzed (Participants) | 28 | 52 | 20
  Week 4 | 47.9241 (45.6) | 47.0462 (35.7) | 48.3634 (21.3)
  Week 6: number analyzed (Participants) | 28 | 52 | 20
  Week 6 | 36.3003 (286.7) | 41.2410 (183.0) | 52.4876 (38.0)
  Week 8: number analyzed (Participants) | 28 | 52 | 20
  Week 8 | 21.9292 (621.4) | 39.9282 (243.7) | 33.4139 (69.0)
  Week 12: number analyzed (Participants) | 26 | 50 | 20
  Week 12 | 16.1907 (300.7) | 46.9934 (189.3) | 23.8437 (105.9)
  Week 16: number analyzed (Participants) | 26 | 51 | 20
  Week 16 | 14.5995 (405.5) | 48.3156 (183.8) | 18.1204 (381.8)
  Week 24: number analyzed (Participants) | 21 | 49 | 20
  Week 24 | 26.2596 (52.8) | 51.6911 (118.2) | 7.7206 (1747.5)
  Week 32: number analyzed (Participants) | 20 | 49 | 19
  Week 32 | 26.9398 (48.8) | 44.5749 (177.2) | 8.4148 (1245.6)
  Week 40: number analyzed (Participants) | 19 | 48 | 17
  Week 40 | 22.2790 (68.3) | 50.9685 (53.3) | 16.7013 (231.1)
  Week 52: number analyzed (Participants) | 19 | 45 | 17
  Week 52 | 20.4541 (90.8) | 54.1341 (43.4) | 15.9290 (149.1)
  Early Withdrawal: number analyzed (Participants) | 4 | 6 | 0
  Early Withdrawal | 0.8342 (5520.7) | 0.6115 (49802.8) |
  Safety Follow-Up: number analyzed (Participants) | 27 | 53 | 20
  Safety Follow-Up | 0.1739 (757.5) | 0.3760 (1460.3) | 0.1407 (714.5)

7. Secondary Outcome: Percentage of Participants With Positive Anti-Certolizumab Pegol-antibody Levels in Plasma
Description: A pre-anti-drug (CZP) antibody (ADA) positive subject was defined as having a confirmed positive sample at Baseline. A pre-ADA negative subject was defined as having a Screening below the cut point (BCP) sample, or a screening above the cut point (ACP) sample, but not confirmed positive at Baseline.
  A treatment-emergent ADA positive subject was defined as either 1) pre-ADA negative subjects having at least 1 ADA confirmed positive sample or 2) pre-ADA positive subjects with at least 1 sample with greater then or equal to (>=) 1.67-fold increase from Baseline on CZP treatment.
Time Frame: Blood samples will be collected at Baseline (Week 0) and at Weeks 2, 4, 6, 8, 12, 16, 24, 32, 40, 52, 60
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | CZP 200 mg Q2W/CZP 200 mg Q2W (PK-PPS) | CZP 400 mg Q2W/CZP 400 mg Q2W (PK-PPS) | CZP 200 mg Q2W/CZP 400 mg Q4W (PK-PPS)
Number analyzed (Participants) | 28 | 53 | 20
percentage of participants | 100 | 96.2 | 90.0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from Baseline (Week 0) until the Safety Follow-up Visit (Week 60).
Description: Until Week 16 (Initial Period), there were 26 pts of PBO, 48 pts of CZP 200 mg, 53 pts of CZP 400 mg, but the safety set up to Week 52 was Escape Arm after Week 16, and CZP was administered. Therefore, Combined Initial and Maintenance Period is evaluated by the number of pts actually administered according to the dose of CZP.
Groups:
- Placebo (SS): This arm consisted of participants who received at least one dose of Placebo subcutaneous (sc) injection every two weeks (Q2W) during the study. Participants formed the Safety Set (SS).
- CZP 200mg Q2W (SS): This arm consisted of participants who received at least one dose of Certolizumab Pegol (CZP) subcutaneous (sc) injection 200 mg every two weeks (Q2W) during the study. Participants formed the SS.
- CZP 400mg Q4W (SS): This arm consisted of participants who received at least one dose of Certolizumab Pegol (CZP) subcutaneous (sc) injection 400 mg every four weeks (Q4W) during the study. Participants formed the SS.
- CZP 200 mg Q2W + CZP 400 mg Q4W (SS): This arm consisted of participants who received at least one dose of Certolizumab Pegol (CZP) subcutaneous (sc) injection 200 mg every two weeks (Q2W) and at least one dose of Certolizumab Pegol (CZP) subcutaneous (sc) injection 400 mg every four weeks (Q4W) during the study. Participants formed the SS.
- CZP 400 mg Q2W (SS): This arm consisted of participants who received at least one dose of Certolizumab Pegol (CZP) subcutaneous (sc) injection 400 mg every two weeks (Q2W) during the study. Participants formed the SS.
- All CZP (SS): This arm consisted of participants who received at least one dose of Certolizumab Pegol (CZP) subcutaneous (sc) injection regardless of the dose during the study. Participants formed the SS.
Arm/Group | Placebo (SS) | CZP 200mg Q2W (SS) | CZP 400mg Q4W (SS) | CZP 200 mg Q2W + CZP 400 mg Q4W (SS) | CZP 400 mg Q2W (SS) | All CZP (SS)
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/72 | 0/20 | 0/72 | 0/64 | 0/122
Serious Adverse Events (participants affected / at risk) | 1/26 | 2/72 | 0/20 | 2/72 | 6/64 | 8/122
Other Adverse Events (participants affected / at risk) | 17/26 | 41/72 | 15/20 | 48/72 | 45/64 | 91/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (SS) (N=26) | CZP 200mg Q2W (SS) (N=72) | CZP 400mg Q4W (SS) (N=20) | CZP 200 mg Q2W + CZP 400 mg Q4W (SS) (N=72) | CZP 400 mg Q2W (SS) (N=64) | All CZP (SS) (N=122)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dental cyst (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Latent tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (SS) (N=26) | CZP 200mg Q2W (SS) (N=72) | CZP 400mg Q4W (SS) (N=20) | CZP 200 mg Q2W + CZP 400 mg Q4W (SS) (N=72) | CZP 400 mg Q2W (SS) (N=64) | All CZP (SS) (N=122)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 1 (1) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 4 (4)
Folliculitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 3 (4) | 6 (7)
Myringitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 3 (4) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 4 (4)
Dermatophytosis of nail (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 5 (5)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Tinea versicolour (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 6 (8) | 23 (24) | 6 (6) | 25 (30) | 28 (48) | 53 (78)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cell marker increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 2 (2) | 4 (5) | 3 (4) | 7 (9)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 4 (6) | 7 (10)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (5) | 0 (0) | 4 (5) | 3 (4) | 7 (9)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (7) | 0 (0) | 5 (7) | 4 (4) | 9 (11)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 6 (6)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (3) | 0 (0) | 2 (3) | 1 (1) | 3 (4)
Psoriasis (Skin and subcutaneous tissue disorders) | 6 (6) | 8 (8) | 0 (0) | 8 (8) | 5 (5) | 13 (13)
Essential hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-01-25): https://cdn.clinicaltrials.gov/large-docs/17/NCT03051217/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/17/NCT03051217/SAP_001.pdf